CLINICAL TRIAL: NCT05289349
Title: Postoperative Effects of Propofol or Sevoflurane Anesthesia in Egyptian Patients
Brief Title: Propofol or Sevoflurane Anesthesia in Egyptian Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehab Werida (Other)
Responsible Party: Sponsor-Investigator, Rehab Werida, Principal Investigator, Damanhour University
Organization: Damanhour University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Propofol/Sevofluran Anesthesia
Record Dates: First submitted 2022-03-13; First posted 2022-03-21 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Anesthesia
Keywords: Postoperative Effects.; Propofol; Sevoflurane; Anesthesia
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Intervention Model Description: prospective, randomized (1:1), double blind clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (P) for propofol (Active Comparator): propofol 6 mg/kg/h in group P
  Interventions: Drug: Propofol
- group (S) for sevoflurane. (Active Comparator): sevoflurane 1.0-1.5 minimum alveolar concentration (MAC) in group S.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — Propofol (2 mg/kg) for induction of anesthesia , and ( 6 mg/kg/h) for maintenance of anesthesia
  Arms: group (P) for propofol
Drug: Sevoflurane — Sevoflurane 1.0-1.5 minimum alveolar concentration (MAC)
  Other Names: Sevoflurane inhalant product
  Arms: group (S) for sevoflurane.

SUMMARY:
The proposed research in this application will investigate postoperative cognitive function, pain index, inflammatory response, and oxidative stress effects of propofol versus sevoflurane anesthetic drugs in patients undergoing elective, non-cardiac abdominal operations under general anesthesia to investigate which of them will significantly maintain better cognitive function, decrease the pain index, inflammatory reaction, and oxidative stress, improve outcome, shorten the postoperative recovery time and reduce length of hospital stay, and consequently the cost of hospital stay.

DETAILED DESCRIPTION:
1. Ethical committee approval will be obtained from Ethics committee of Faculty of Pharmacy, Damanhour University.
2. Ethical committee approval will be obtained from Ethics committee of General Organization for Teaching Hospitals and Institutes.
3. About 44 patients who are candidate for elective, non-cardiac abdominal surgery under general anesthesia with either propofol infusion or sevoflurane inhalation, will be recruited from Damanhour Teaching Hospital, General Organization for Teaching Hospitals and Institutes.
4. All participants should agree to take part in this clinical study and will provide informed consent.
5. Demographic data; age (year), sex (female/male), weight (kg), height (cm), BMI (kg/m2) will be collected.
6. ASA physical status will be recorded.
7. Venous blood samples (5 ml will be collected by a sterile syringe then placed in a suitable sterile tube to be centrifuged, the serum will be reserved and stored at -80°C until the analysis) before, and 1 hour after operation for evaluating cognitive function by analyses of Neuron Specific Enolase (NSE, µg/L) and (S100-β protein, pg/mL) and for determining inflammatory response by measuring Matrix Metallo-Proteinase-9 (MMP-9, ng/mL), and effect of these anesthetic drugs on oxidative stress by measuring Super Oxide Dismutase (SOD, U/L).
8. Cognitive function scale: Mini-Mental State Examination (MMSE scale, if decreased more than 2 points from before operation indicate that the cognitive function of patients are declined) and pain index: Numerical Pain Rating scale (NPRS) (a scale from 0-10, where 0 = no pain and 10 = maximum worst pain) will be performed on all patients before, 1 hour, and 24 hours after operation.
9. Heart rate (beat/min), oxygen saturation (%), and non-invasive blood pressure (mmHg) (systolic, diastolic, mean) will be recorded before and after operation.

10 Anesthesia duration (min) (the time from induction of anesthesia till stoppage of anesthesia) and operative duration (min) (the time from skin incision till skin closure) will be recorded.

11. Time to emerge from anesthesia (min) (the time from stopping the use of anesthetics to patients relatively clearly answering the doctor's questions) will be recorded.

12. The incidence of any perioperative adverse effects will be recorded as; tachycardia, bradycardia, hypertension, hypotension, nausea, vomiting, hypoxia, and bleeding.

* Study design: This is a prospective, randomized (1:1), clinical trial, will be carried out on 44 patients who are candidate for elective, major, non-cardiac operations under general anesthesia.
* Patients will be randomly allocated into two equal groups (22 patients each); group (P) for propofol and group (S) for sevoflurane.
* The day before the operation, patients will be taught to measure postoperative pain based on the NPRS. Patients will be fasting for 6-8 h for a solid meal and 2 hours for clear fluid before the operation.
* On arrival to the operating room, a peripheral IV cannula will be secured and standard monitoring using an electrocardiogram, pulse oximetry, and non-invasive blood pressure will be applied.
* After preoxygenation with 100% oxygen for 3 min, general anesthesia will be induced using IV propofol (2 mg/kg) and IV fentanyl (1 μg/kg), and IV atracurium (0.5 mg/kg) will be given to facilitate tracheal intubation.
* Lungs will be ventilated using volume-controlled ventilation and the tidal volume and ventilation rate will be adjusted to maintain end-tidal carbon dioxide at 35-45 mmHg.
* Anesthesia will be maintained with either total intravenous anesthesia (TIVA) with propofol 6 mg/kg/h in group P or sevoflurane 1.0-1.5 minimum alveolar concentration (MAC) in group S.
* Continuous infusion of IV atracurium (0.3 mg/kg/h), and IV fentanyl (0.5 ug/kg/h) till the end of surgery.
* Thirty minutes before the end of the surgery all patients will be given IV paracetamol (15 mg/kg) for postoperative pain management.
* At the end of the surgery, either TIVA pump or the inhalational anesthetic vaporizer will be turned off and the muscle relaxant will be reversed by giving IV neostigmine (0.04 mg/kg) plus IV atropine (0.02 mg/kg).
* The patient will be extubated and transferred to the post-anesthesia care unit.
* All data and study outcomes will be recorded by a researcher who is blinded to group assignment.
* The primary outcome is the measure postoperative cognitive function by NSE.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will be candidates for elective, major, non-cardiac abdominal operations under general anesthesia with propofol or sevoflurane.
2. Patients aged from 21 and older, of either sex.
3. Patients with body mass index (BMI) 25 to 35 kg/m².
4. Patients belong to the American Society of Anesthesiologist (ASA) physical status I or II.
5. Patients should have basically normal preoperative laboratory investigations.

Exclusion Criteria:

1. Patients with mini-mental state examination (MMSE) score <24 points.
2. Patients with significant cardiovascular, cerebrovascular, respiratory, liver, renal, endocrine, blood, or immune diseases.
3. Patients with visual or auditory disease, infection, chronic inflammation, disturbance of consciousness, cognitive impairment, or dementia.
4. Patients who are on long-term use of sedatives or steroids.
5. Alcohol or drug abuse.
6. Allergy to any drug will be used in this study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Neuron Specific Enolase (NSE, µg/L) | 1 hour after operation
  Venous blood Level
S100-β protein, pg/mL | 1 hour after operation
  Venous blood Level
Matrix Metallo-Proteinase-9 (MMP-9, ng/mL) | 1 hour after operation
  Venous blood Level
Super Oxide Dismutase (SOD, U/L) | 1 hour after operation
  Venous blood Level

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass Prof., Study Chair — Damanhour University; Amira Kassem, Ph.D, Principal Investigator — Damanhour University; Ahmed Shaat, Ph.D., Principal Investigator — Damanhour Teaching Hospital; Heba Elwan, Principal Investigator — Damanhour University; Ahmad Salahuddin, Ph.D, Principal Investigator — Damanhour University
Locations (1):
- Damanhour Teaching Hospital, General Organization for Teaching Hospitals and Institutes., Damanhūr, Elbehairah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caza N, Taha R, Qi Y, Blaise G. The effects of surgery and anesthesia on memory and cognition. Prog Brain Res. 2008;169:409-22. doi: 10.1016/S0079-6123(07)00026-X. PMID 18394490
- [Background] Tian HT, Duan XH, Yang YF, Wang Y, Bai QL, Zhang X. Effects of propofol or sevoflurane anesthesia on the perioperative inflammatory response, pulmonary function and cognitive function in patients receiving lung cancer resection. Eur Rev Med Pharmacol Sci. 2017 Dec;21(23):5515-5522. doi: 10.26355/eurrev_201712_13943. PMID 29243798
- [Background] Zhao Y, Zhang H. Propofol and sevoflurane combined with remifentanil on the pain index, inflammatory factors and postoperative cognitive function of spine fracture patients. Exp Ther Med. 2018 Apr;15(4):3775-3780. doi: 10.3892/etm.2018.5898. Epub 2018 Feb 27. PMID 29563982